CLINICAL TRIAL: NCT02715076
Title: The Effects of Ambient Temperature and Forced-air Warming on Intraoperative Core Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Lijian Pei, Associate Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: ZS-878
Record Dates: First submitted 2016-02-29; First posted 2016-03-22 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Major Surgery Under General Anesthesia
Keywords: Thoracic Surgery; Thoracic surgery, Video assisted; Open Abdominal Surgery; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ambient Temp 19°C & Passive Insulation (Experimental): Ambient Temperature 19°C and Passive Insulation: patients assigned to passive insulation will be covered as usual with a cotton gown and single layer of cloth surgical draping.
  Interventions: Other: Ambient Temperature 19°C; Other: Passive insulation
- Ambient Temp 19°C & Forced-air Warming (Experimental): Ambient Temperature 19°C and Forced-air Warming: patients assigned to forced-air warming will also be covered with a gown and surgical drapes, but a forced-air cover (Bair hugger 63500, 3M) will be inserted between the gown and the skin surface.
  Interventions: Other: Ambient Temperature 19°C; Device: Forced-air cover (Bair hugger 63500, 3M)
- Ambient Temp 21°C & Passive Insulation (Experimental): Ambient Temperature 21°C and Passive Insulation: patients assigned to passive insulation will be covered as usual with a cotton gown and single layer of cloth surgical draping.
  Interventions: Other: Ambient Temperature 21°C; Other: Passive insulation
- Ambient Temp 21°C & Forced-air Warming (Experimental): Ambient Temperature 21°C and Forced-air Warming: patients assigned to forced-air warming will also be covered with a gown and surgical drapes, but a forced-air cover (Bair hugger 63500, 3M) will be inserted between the gown and the skin surface.
  Interventions: Other: Ambient Temperature 21°C; Device: Forced-air cover (Bair hugger 63500, 3M)
- Ambient Temp 23°C & Passive Insulation (Experimental): Ambient Temperature 23°C and Passive Insulation: patients assigned to passive insulation will be covered as usual with a cotton gown and single layer of cloth surgical draping.
  Interventions: Other: Ambient Temperature 23°C; Other: Passive insulation
- Ambient Temp 23°C & Forced-air Warming (Experimental): Ambient Temperature 23°C and Forced-air Warming: patients assigned to forced-air warming will also be covered with a gown and surgical drapes, but a forced-air cover (Bair hugger 63500, 3M) will be inserted between the gown and the skin surface.
  Interventions: Other: Ambient Temperature 23°C; Device: Forced-air cover (Bair hugger 63500, 3M)

INTERVENTIONS:
Other: Ambient Temperature 19°C — Ambient Temperature 19°C
  Arms: Ambient Temp 19°C & Forced-air Warming; Ambient Temp 19°C & Passive Insulation
Other: Ambient Temperature 21°C — Ambient Temperature 21°C
  Arms: Ambient Temp 21°C & Forced-air Warming; Ambient Temp 21°C & Passive Insulation
Other: Ambient Temperature 23°C — Ambient Temperature 23°C
  Arms: Ambient Temp 23°C & Forced-air Warming; Ambient Temp 23°C & Passive Insulation
Device: Forced-air cover (Bair hugger 63500, 3M) — Patients assigned to forced-air warming will also be covered with a gown and surgical drapes, but a forced-air cover (Bair hugger 63500, 3M) will be inserted between the gown and the skin surface.
  Arms: Ambient Temp 19°C & Forced-air Warming; Ambient Temp 21°C & Forced-air Warming; Ambient Temp 23°C & Forced-air Warming
Other: Passive insulation — Patients assigned to passive insulation will be covered as usual with a cotton gown and single layer of cloth surgical draping.
  Arms: Ambient Temp 19°C & Passive Insulation; Ambient Temp 21°C & Passive Insulation; Ambient Temp 23°C & Passive Insulation

SUMMARY:
The purpose of this study is to determine:

1. the effect of ambient temperature on the rate of core temperature change from 1 to 3 hours after induction of anesthesia (linear phase of the hypothermia curve) in major operations lasting at least a couple of hours and
2. whether the relationship between ambient temperature and rate of core temperature change is different for patients who are or are not warmed with forced-air.

DETAILED DESCRIPTION:
Each patient will be randomly assigned to ambient temperature of 19°C, 21°C, or 23°C. Using a factorial approach, patients will also be randomly assigned to passive insulation or forced-air warming, stratified by the three types of surgery listed below. Group allocation will be based on computer generated codes (randomly permuted block sizes) prepared by Department of OUTCOMES RESEARCH statisticians using SAS statistical software. Allocation of consented patients to designated ambient temperature and forced-air vs. passive insulation will be via a web site that will be accessed by investigators in Bejing about 90 minutes before surgery.

Patients assigned to passive insulation will be covered as usual with a cotton gown and single layer of cloth surgical draping. Patients assigned to forced-air warming will also be covered with a gown and surgical drapes, but a forced-air cover (Bair hugger 63500, 3M) will be inserted between the gown and the skin surface. A lower-body cover (about 91 by 221 cm) will be positioned so the lower end of the forced-air segments extend from the ankles upward for the entire length of the cover in thoracic and abdominal cases. The cover's foot drape will extend over the feet, and in turn be covered by the surgical drape. An upper-body forced-air cover will similarly be applied for patients having hip arthroplasties. The forced-air cover will be connected to a Bair Hugger blower and #635 covers set to "high" (≈43°C).

Ambient temperature will be adjusted to the designated temperature about an hour before a patient enters the operating room and adjusted as necessary to maintain the designated temperature throughout surgery. General anesthesia will be induced as per usual clinical routine. Neuraxial (epidural or spinal) and other regional blocks are permitted.

Any patients whose core temperature decreases to less than 34.5°C will be actively warmed with forced air and the ambient temperature increases to the extent practical.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for major open thoracic surgery or video assist thoracic surgery or major abdominal surgery under general anesthesia expected to last at least two hours

Exclusion Criteria:

* Special risk for bleeding or myocardial infarction (as determined by the attending anesthesiologist)
* Patients who would otherwise have been actively warmed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LiJian Pei, MD, Principal Investigator — Associate Prof. of Dept. of Anesthesiology, PUMCH; Yuguang Huang, MD, Study Chair — Chair of Dept. of Anesthesiology, PUMCH; Daniel I Sessler, MD, Study Director — Chair of Dept. of Outcomes Research, Anesthesiology Institute, Cleveland Clinic
Locations (1):
- Dept. of Anesthesiology, PUMCH, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hynson JM, Sessler DI. Intraoperative warming therapies: a comparison of three devices. J Clin Anesth. 1992 May-Jun;4(3):194-9. doi: 10.1016/0952-8180(92)90064-8. PMID 1610573
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Lenhardt R, Marker E, Goll V, Tschernich H, Kurz A, Sessler DI, Narzt E, Lackner F. Mild intraoperative hypothermia prolongs postanesthetic recovery. Anesthesiology. 1997 Dec;87(6):1318-23. doi: 10.1097/00000542-199712000-00009. PMID 9416715
- [Background] Kurz A, Sessler DI, Narzt E, Bekar A, Lenhardt R, Huemer G, Lackner F. Postoperative hemodynamic and thermoregulatory consequences of intraoperative core hypothermia. J Clin Anesth. 1995 Aug;7(5):359-66. doi: 10.1016/0952-8180(95)00028-g. PMID 7576669
- [Background] Matsukawa T, Sessler DI, Christensen R, Ozaki M, Schroeder M. Heat flow and distribution during epidural anesthesia. Anesthesiology. 1995 Nov;83(5):961-7. doi: 10.1097/00000542-199511000-00008. PMID 7486181
- [Background] Matsukawa T, Sessler DI, Sessler AM, Schroeder M, Ozaki M, Kurz A, Cheng C. Heat flow and distribution during induction of general anesthesia. Anesthesiology. 1995 Mar;82(3):662-73. doi: 10.1097/00000542-199503000-00008. PMID 7879935
- [Background] Hynson JM, Sessler DI, Moayeri A, McGuire J, Schroeder M. The effects of preinduction warming on temperature and blood pressure during propofol/nitrous oxide anesthesia. Anesthesiology. 1993 Aug;79(2):219-28, discussion 21A-22A. doi: 10.1097/00000542-199308000-00005. PMID 8342834
- [Background] Camus Y, Delva E, Sessler DI, Lienhart A. Pre-induction skin-surface warming minimizes intraoperative core hypothermia. J Clin Anesth. 1995 Aug;7(5):384-8. doi: 10.1016/0952-8180(95)00051-i. PMID 7576673
- [Background] Kurz A, Sessler DI, Christensen R, Dechert M. Heat balance and distribution during the core-temperature plateau in anesthetized humans. Anesthesiology. 1995 Sep;83(3):491-9. doi: 10.1097/00000542-199509000-00007. PMID 7661349
- [Background] Roe CF. Effect of bowel exposure on body temperature during surgical operations. Am J Surg. 1971 Jul;122(1):13-5. doi: 10.1016/0002-9610(71)90338-2. No abstract available. PMID 5091847
- [Background] Rajek A, Greif R, Sessler DI, Baumgardner J, Laciny S, Bastanmehr H. Core cooling by central venous infusion of ice-cold (4 degrees C and 20 degrees C) fluid: isolation of core and peripheral thermal compartments. Anesthesiology. 2000 Sep;93(3):629-37. doi: 10.1097/00000542-200009000-00010. PMID 10969294
- [Background] Sessler DI, McGuire J, Moayeri A, Hynson J. Isoflurane-induced vasodilation minimally increases cutaneous heat loss. Anesthesiology. 1991 Feb;74(2):226-32. doi: 10.1097/00000542-199102000-00006. PMID 1990897
- [Background] Sessler DI, McGuire J, Sessler AM. Perioperative thermal insulation. Anesthesiology. 1991 May;74(5):875-9. doi: 10.1097/00000542-199105000-00012. PMID 2021204
- [Background] Sessler DI, Moayeri A. Skin-surface warming: heat flux and central temperature. Anesthesiology. 1990 Aug;73(2):218-24. PMID 2382847
- [Background] Giesbrecht GG, Ducharme MB, McGuire JP. Comparison of forced-air patient warming systems for perioperative use. Anesthesiology. 1994 Mar;80(3):671-9. doi: 10.1097/00000542-199403000-00026. PMID 8141463
- [Background] Morris RH. Influence of ambient temperature on patient temperature during intraabdominal surgery. Ann Surg. 1971 Feb;173(2):230-3. doi: 10.1097/00000658-197102000-00008. No abstract available. PMID 5100096
- [Background] Morris RH. Operating room temperature and the anesthetized, paralyzed patient. Arch Surg. 1971 Feb;102(2):95-7. doi: 10.1001/archsurg.1971.01350020005002. No abstract available. PMID 4250862
- [Background] Morris RH, Wilkey BR. The effects of ambient temperature on patient temperature during surgery not involving body cavities. Anesthesiology. 1970 Feb;32(2):102-7. doi: 10.1097/00000542-197002000-00003. No abstract available. PMID 5414287
- [Background] Wang CS, Chen CL, Huang CJ, Cheng KW, Chen KH, Wang CC, Concejero AM, Cheng YF, Huang TL, Wang SH, Lin CC, Liu YW, Yong CC, Yang CH, Jawan B. Effects of different operating room temperatures on the body temperature undergoing live liver donor hepatectomy. Transplant Proc. 2008 Oct;40(8):2463-5. doi: 10.1016/j.transproceed.2008.07.077. PMID 18929769
- [Background] Tander B, Baris S, Karakaya D, Ariturk E, Rizalar R, Bernay F. Risk factors influencing inadvertent hypothermia in infants and neonates during anesthesia. Paediatr Anaesth. 2005 Jul;15(7):574-9. doi: 10.1111/j.1460-9592.2005.01504.x. PMID 15960641
- [Background] Ozer AB, Tosun F, Demirel I, Unlu S, Bayar MK, Erhan OL. The effects of anesthetic technique and ambient temperature on thermoregulation in lower extremity surgery. J Anesth. 2013 Aug;27(4):528-34. doi: 10.1007/s00540-013-1555-2. Epub 2013 Jan 23. PMID 23340983
- [Background] Cheng KW, Wang CH, Chen CL, Jawan B, Wang CC, Concejero AM, Wang SH, Liu YW, Yong CC, Yang CH, Huang CJ. Decreased fresh gas flow cannot compensate for an increased operating room temperature in maintaining body temperature during donor hepatectomy for living liver donor hepatectomy. Transplant Proc. 2010 Apr;42(3):703-4. doi: 10.1016/j.transproceed.2010.02.065. PMID 20430151
- [Background] Frank SM, Beattie C, Christopherson R, Norris EJ, Rock P, Parker S, Kimball AW Jr. Epidural versus general anesthesia, ambient operating room temperature, and patient age as predictors of inadvertent hypothermia. Anesthesiology. 1992 Aug;77(2):252-7. doi: 10.1097/00000542-199208000-00005. PMID 1642343
- [Derived] Sun C, Gao H, Zhang Y, Pei L, Huang Y. Risk Stratification for Organ/Space Surgical Site Infection in Advanced Digestive System Cancer. Front Oncol. 2021 Nov 9;11:705335. doi: 10.3389/fonc.2021.705335. eCollection 2021. PMID 34858805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ambient Temp 19°C & Passive Insulation | Ambient Temp 19°C & Forced-air Warming | Ambient Temp 21°C & Passive Insulation | Ambient Temp 21°C & Forced-air Warming | Ambient Temp 23°C & Passive Insulation | Ambient Temp 23°C & Forced-air Warming
Started | 48 | 50 | 49 | 50 | 47 | 48
Completed | 48 | 50 | 49 | 50 | 47 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambient Temp 19°C & Passive Insulation | Ambient Temp 19°C & Forced-air Warming | Ambient Temp 21°C & Passive Insulation | Ambient Temp 21°C & Forced-air Warming | Ambient Temp 23°C & Passive Insulation | Ambient Temp 23°C & Forced-air Warming | Total
Number analyzed (Participants) | 48 | 50 | 49 | 50 | 47 | 48 | 292
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 54 (12) | 54 (13) | 57 (11) | 57 (11) | 54 (12) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 27 | 24 | 18 | 22 | 24 | 144
  Male | 19 | 23 | 25 | 32 | 25 | 24 | 148

OUTCOME MEASURES:

1. Primary Outcome: Rate of Core Temperature Change
Description: Rate of core temperature change from 1 to 3 hours after induction of anesthesia (°C/hour ) linear mixed-effects model to assess the effects of ambient temperature, forced-air warming and their interaction on the rate of core temperature change during 1 to 3h after induction
Time Frame: from 1 to 3 hours after induction of anesthesia
Population: We plotted the mean core temperatures at 10-minute intervals. The trend of core temperature in each of the six groups between 1 to 3 hours was roughly linear. We thus used the slope (change in °C/hour) to characterize the rate sat which intraoperative core temperature changed.
Measure: Mean (Standard Deviation); unit: degree C
Arm/Group | Ambient Temp 19°C & Passive Insulation | Ambient Temp 19°C & Forced-air Warming | Ambient Temp 21°C & Passive Insulation | Ambient Temp 21°C & Forced-air Warming | Ambient Temp 23°C & Passive Insulation | Ambient Temp 23°C & Forced-air Warming
Number analyzed (Participants) | 48 | 50 | 49 | 50 | 47 | 48
degree C | -0.18 (0.03) | 0.05 (0.03) | -0.06 (0.03) | 0.07 (0.03) | -0.05 (0.03) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Ambient Temp 19°C & Passive Insulation vs Ambient Temp 19°C & Forced-air Warming vs Ambient Temp 21°C & Passive Insulation vs Ambient Temp 21°C & Forced-air Warming vs Ambient Temp 23°C & Passive Insulation vs Ambient Temp 23°C & Forced-air Warming; Test type: Other; p < 0.05, mixed-effects model

ADVERSE EVENTS:
Time Frame: 1 month postoperatively
Description: AKI, SSI
Arm/Group | Ambient Temp 19°C & Passive Insulation | Ambient Temp 19°C & Forced-air Warming | Ambient Temp 21°C & Passive Insulation | Ambient Temp 21°C & Forced-air Warming | Ambient Temp 23°C & Passive Insulation | Ambient Temp 23°C & Forced-air Warming
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/50 | 0/49 | 0/50 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/49 | 0/50 | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 1/48 | 1/50 | 1/49 | 1/50 | 1/47 | 2/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ambient Temp 19°C & Passive Insulation (N=48) | Ambient Temp 19°C & Forced-air Warming (N=50) | Ambient Temp 21°C & Passive Insulation (N=49) | Ambient Temp 21°C & Forced-air Warming (N=50) | Ambient Temp 23°C & Passive Insulation (N=47) | Ambient Temp 23°C & Forced-air Warming (N=48)
surgical site infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No